CLINICAL TRIAL: NCT01807416
Title: Bone Dimensional Changes at Different Implant-to-abutment Connections: a 1-year Clinical and Radiological Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Proed, Torino, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02.2013.Piemonte.PROED
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Osseointegrated Implant, Bone level
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- standard platform , standard abutment (Active Comparator): implant insertion and abutment connection Osseointegrated implants with regular collar connected to standard designed prosthetic abutments
  Interventions: Procedure: implant insertion and abutment connection
- standard platform, flat abutment (Active Comparator): implant insertion and abutment connection Osseointegrated implants with regular collar connected to flat designed prosthetic abutments
  Interventions: Procedure: implant insertion and abutment connection
- switching platform, standard abutment (Active Comparator): implant insertion and abutment connection Osseointegrated implants with switched platform collar connected to standard designed prosthetic abutments
  Interventions: Procedure: implant insertion and abutment connection
- switching platform, flat abutment (Active Comparator): implant insertion and abutment connection Osseointegrated implants with switched platform collar connected to flat designed prosthetic abutments
  Interventions: Procedure: implant insertion and abutment connection

INTERVENTIONS:
Procedure: implant insertion and abutment connection — After implant insertion (standard platform or switching platform) the titanium abutment (standard or flat) will be connected

SUMMARY:
Aim of the present study will be to evaluate if the platform switching and the flat abutment can modify the peri-implant marginal bone remodelling. A clinical assessment of the soft tissues will also be provided.

80 consecutively inserted dental implants will be included in this study. Maxillary and mandibular implants will be considered, both in frontal and posterior area. After 6 to 12 weeks, the definitive prosthetic abutment will be screwed and the temporary crown cemented. After 2 more months, the definitive porcelain crown will be delivered. The final outcomes will be collected after 1 year from implant insertion.

Data will refer to the following timing:

T0= implant installation T1= temporary crown cementation T2= definitive crown cementation T3= 1 year follow-up The 80 implants will be randomly divided into 4 groups of 20 implants each, with different implant/abutment design.

Group 1: Tapered T3 Standard Collar implants + GingiHue abutments Group 2: Tapered T3 Standard Collar implants + Tissuemax IL abutments Group 3: Tapered T3 Prevail implants + GingiHue abutments Group 4: Tapered T3 Prevail implants + Tissuemax IL abutments On x-rays, the mesial and distal Marginal Bone Level will be measured and compared among and between the groups at the 4 different timing.

Pocket Depth and Bleeding on probing (mesial, buccal, distal and lingual) will be measured at T0, T1, T2 and T3. Data will be statistically analyzed.

DETAILED DESCRIPTION:
BACKGROUND:

Platform switching is intended to preserve marginal bone around implants. Studies have shown that implants using an integrated platform switching demonstrate crestal bone loss as low as 0.37mm, and 30 to 50% reduction in crestal bone loss when compared to non-platform switching implants. Recently, a new design titanium abutment (Tissuemax IL) has been proposed to modulate the soft tissue integration around implant supported crowns. A new implant with a hybrid surface (T3) has been recently launched by Biomet 3i, providing both integrated platform switching (Prevail) or non platform switching (Standard Collar).

Aim of the present study will be to evaluate if the platform switching and the Tissuemax abutment can modify the peri-implant marginal bone remodelling. A clinical assessment of the soft tissues will also be provided.

MATERIALS & METHODS:

80 consecutively inserted dental implants will be included in this study. Maxillary and mandibular implants will be considered, both in frontal and posterior area. Implants should be inserted in preexisting adequate bone volume, without the need for any bone augmentation technique. Implants will be inserted with a transmucosal healing (single-stage surgical procedure) with immediate connection of the healing abutment. After 6 to 12 weeks, the definitive prosthetic abutment will be screwed and the temporary crown cemented. After 2 more months, the definitive porcelain crown will be delivered. The final outcomes will be collected after 1 year from implant insertion.

Data will refer to the following timing:

T0= implant installation T1= temporary crown cementation T2= definitive crown cementation T3= 1 year follow-up The 80 implants will be randomly divided into 4 groups of 20 implants each, with different implant/abutment design.

Group 1: Tapered T3 Standard Collar implants + GingiHue abutments Group 2: Tapered T3 Standard Collar implants + Tissuemax IL abutments Group 3: Tapered T3 Prevail implants + GingiHue abutments Group 4: Tapered T3 Prevail implants + Tissuemax IL abutments The division into the 4 group will be randomized. Standardized intraoral radiograms will be done at T0, T1, T2 and T3. On x-rays, the mesial and distal Marginal Bone Level will be measured and compared among and between the groups at the 4 different timing.

Pocket Depth and Bleeding on probing (mesial, buccal, distal and lingual) will be measured at T0, T1, T2 and T3. Data will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult patients with partial edentulism

Exclusion Criteria:

* Current pregnant patients
* History of malignancy
* History of radiotherapy or chemiotherapy in the last 5 years
* Long term steroidal or antibiotic therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Marginal Bone Level | 1 year after implant installation
  On standardized intraoral radiograms, mesial and distal marginal bone level at implant surface will be measured

SECONDARY OUTCOMES:
Probing Pocket Depth | 1 year after implant installation
  Probing depth measured mesially, buccaly, distally and lingually at implant site
Bleeding on Probing | 1 year after implant installation
  Bleeding on Probing measured mesially, buccaly, distally and lingually at implant site

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Cardaropoli, DDS, Study Director — Proed, Torino, Italy
Locations (1):
- PROED, Institute for Professional Education in Dentistry, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: No